CLINICAL TRIAL: NCT04083144
Title: Deep rTMS and Varenicline for Smoking Cessation: A Pilot Study Exploring the Efficacy of a Combined Treatment Approach
Brief Title: Deep rTMS and Varenicline for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Pfizer (Industry); Brainsway (Industry)
Responsible Party: Principal Investigator, Bernard Le Foll, Head,Translational Addiction Research Laboratory, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 051/2017
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Tobacco Use Disorder; Smoking Cessation
Keywords: smoking cessation; varenicline; deep rTMS; insula; addiction; tobacco use disorder
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Behavior, Addictive | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep rTMS active + Varenicline (Active Comparator): Participants undergoing deep rTMS (active) for 4 weeks (5 sessions/week) along with 12 weeks of varenicline.
  Interventions: Device: Deep Repetitive Transcranial Magnetic Stimulation (Active); Drug: Varenicline
- Deep rTMS sham + Varenicline (Sham Comparator): Participants undergoing deep rTMS (sham) for 4 weeks (5 sessions/week) along with 12 weeks of varenicline.
  Interventions: Device: Deep Repetitive Transcranial Magnetic Stimulation (Sham); Drug: Varenicline

INTERVENTIONS:
Device: Deep Repetitive Transcranial Magnetic Stimulation (Active) — Active deep rTMS (10 Hz) using the H-coil to target the bilateral insula
  Arms: Deep rTMS active + Varenicline
Device: Deep Repetitive Transcranial Magnetic Stimulation (Sham) — Sham deep rTMS using the H-coil. The sham coil is built into the same helmet as the active coil. It mimics the active coil with regards to acoustics and scalp sensations.
  Arms: Deep rTMS sham + Varenicline
Drug: Varenicline — 12 week course treatment of varenicline (0.5 mg/1 mg) using the standard dosage schedule for smoking cessation (Day 1-3: 0.5 mg daily; day 4-7: 0.5 mg twice a day; day 8-end of treatment: 1 mg twice a day).
  Other Names: Champix

SUMMARY:
The purpose of this study is to investigate the effect of deep repetitive transcranial magnetic stimulation (rTMS) using the insula H-coil on smoking outcomes in smokers receiving varenicline. It is hypothesized that active deep rTMS will improve abstinence rates, attenuate craving and reduce cigarette consumption and dependence severity.

DETAILED DESCRIPTION:
This study will be a randomized, double-blind, sham-controlled clinical trial. Nicotine dependent participants will be recruited and randomized tor receive either active or sham rTMS intervention for 4 weeks (5 sessions/week). All participants will receive an open-label treatment of varenicline for 12 weeks and weekly counselling sessions. The aims of the study are:

1. To examine the efficacy of bilateral deep rTMS to the insula on point prevalence smoking abstinence in smokers receiving varenicline treatment.
2. To examine the efficacy of bilateral deep rTMS to the insula on other smoking outcomes such as craving, cigarette smoking and dependence severity.
3. To examine the effect of bilateral deep rTMS to the insula on abstinence at the end of rTMS treatment and at 6-month follow up.

Abstinence will be measured by point prevalence at week 4 and 12 and prolonged continuous abstinence at week 26. This will be confirmed using plasma cotinine levels. All other measures will be done using various questionnaires such as Fagerstrom Test of Nicotine Dependence (FTND), Timeline Follow-Back (TLFB), Minnesota Nicotine Withdrawal Scale (MNWS), and Tiffany Questionnaire of Smoking Urges (T-QSU).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65;
* Nicotine dependent as assessed by Diagnostic and Statistical Manual of Mental Disorders (DSM-V);
* Reported daily cigarette consumption ≥ 10 and expired carbon monoxide (CO) measurement of ≥ 10 ppm;
* Fagerstrom Test of Nicotine Dependence (FTND) ≥ 4;
* Reported motivation to quit within 30 days as assessed using the Contemplation Ladder score of ≥ 7.

Exclusion Criteria:

* Reported smoking abstinence in the 3 months preceding screening visit;
* Current use of other smoking cessation aids;
* Allergy and/or contraindication to varenicline or rTMS;
* Pregnancy, trying to become pregnant or breastfeeding;
* Current or recent history of cardiovascular or cerebrovascular disease and/or current hypertension;
* Current or historical evidence of suicidal behavior;
* Serious current or personal history of medical condition/disease (neurological disorders, brain lesions, multiple sclerosis, head trauma, loss of consciousness, hearing loss, etc.);
* Current, personal history or family history of seizures;
* Cognitive impairment as defined as a Mini Mental State Examination (MMSE) score <24;
* Concomitant use of medication that lowers seizure threshold

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD,PhD,MCFP, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibrahim C, Malik S, Barr MS, Blumberger DM, Daskalakis ZJ, Le Foll B. Insula deep rTMS and varenicline for smoking cessation: A randomized control trial study protocol. Front Pharmacol. 2022 Sep 8;13:969500. doi: 10.3389/fphar.2022.969500. eCollection 2022. PMID 36160428
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — https://www.camh.ca/en/science-and-research

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 participants were enrolled, however, 8 of them were lost to follow up before randomization and therefore were not assigned to any group.
Period: Overall Study
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Started | 24 | 18
Completed | 16 | 15
Not Completed | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline | Total
Number analyzed (Participants) | 24 | 18 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.5) | 46.2 (12.9) | 44.8 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 20 | 10 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Black or African American | 0 | 3 | 3
  White | 19 | 13 | 32
  More than one race | 3 | 2 | 5
Education Level [Count of Participants; unit: Participants]
  Less than grade 8 | 1 | 1 | 2
  Highschool | 8 | 1 | 9
  College/University/Grad School | 15 | 16 | 31
Education Years [Mean (Standard Deviation); unit: years] | 14.8 (3.6) | 14.5 (2.8) | 14.7 (3.05)
Employment Status [Count of Participants; unit: Participants]
  Employed | 15 | 11 | 26
  Unemployed | 6 | 5 | 11
  Retired | 3 | 2 | 5
Housing [Count of Participants; unit: Participants]
  House | 7 | 7 | 14
  Apartment | 15 | 11 | 26
  Condo | 2 | 0 | 2
Income [Count of Participants; unit: Participants]
  <19,999 | 7 | 2 | 9
  20,000-49,999 | 9 | 10 | 19
  50,000-74,999 | 4 | 4 | 8
  >75,000 | 4 | 2 | 6
Marital Status [Count of Participants; unit: Participants]
  Married/Common Law | 6 | 5 | 11
  Separated/Divorced/Annulled | 6 | 4 | 10
  Never Married | 12 | 9 | 21
Fagerström Test for Nicotine Dependence [Mean (Standard Deviation); unit: Score out of 10] — Higher score = higher nicotine dependence severity Score 0-10
  Score out of 10 | 5.6 (1.5) | 6.3 (1.4) | 5.9 (1.47)
Mini-mental state examination [Mean (Standard Deviation); unit: Score out of 30] — Lower score = cognitive impairment Score 0-30
  Score out of 30 | 28.5 (1.5) | 28.4 (1.5) | 28.5 (1.4)
Smoking Contemplation Ladder [Mean (Standard Deviation); unit: Score out of 10] | 9 (1) | 9 (1) | 9 (1)
CO Measurement [Mean (Standard Deviation); unit: ppm] | 24.7 (13.9) | 24.3 (11.3) | 24.5 (11.9)
Cigarettes/day [Mean (Standard Deviation); unit: Cigarettes/day] — The number of cigarettes smoked per day over the past 30 days
  Cigarettes/day | 16.9 (5.3) | 19.4 (1.3) | 18.0 (4.8)
Alcoholic Drinks/day [Mean (Standard Deviation); unit: Drinks/day] — The number of alcoholic drinks consumed per day over the past 30 days
  Drinks/day | 1.1 (1.7) | 1.3 (1.6) | 1.2 (1.6)
Nicotine Metabolite Ratio [Mean (Standard Deviation); unit: Ratio 0-1] — The ratio of 3'hydroxycotinine [3HC]/cotinine
  A low ratio indicates slow nicotine metabolism and a high ratio indicates fast nicotine metabolism. There is no clear cutoff of slow vs. fast metabolizer as it depends on the population studied and the methods used.
  Ratio 0-1 | 0.50 (0.3) | 0.55 (0.22) | 0.52 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Point Prevalence Abstinence at the End of 12 Weeks
Description: Measured by self-report of smoking abstinence in the past 7 days and confirmed using plasma cotinine measurement.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 17 | 15
Participants
  Abstinent | 12 | 6
  Non-abstinent | 5 | 9

2. Secondary Outcome: Fagerstrom Test For Nicotine Dependence (FTND) Score
Description: This will be used to assess physical dependence severity in participants. It is a 6 item scale and total scores can range from 0-10. A higher score indicates more severe nicotine dependence.
Time Frame: 26 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 24 | 18
score on a scale | 0.636 (0.447) | 1.468 (0.47)
Statistical Analysis 1: Comparison: Deep rTMS Active + Varenicline vs Deep rTMS Sham + Varenicline; Test type: Superiority; p = 0.98, Mixed Models Analysis; η2 = 0.01

3. Secondary Outcome: Expired CO Measurements
Description: This will be used as a biological confirmation of recent smoking.
Time Frame: 26 weeks
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 24 | 18
ppm | 8.457 (2.5) | 8.124 (2.624)
Statistical Analysis 1: Comparison: Deep rTMS Active + Varenicline vs Deep rTMS Sham + Varenicline; Test type: Superiority; p = 0.76, Mixed Models Analysis; η2 = 0.16

4. Secondary Outcome: Cigarettes Per Day (TLFB)
Description: Self-reported measure of cigarette consumption.
Time Frame: 26 weeks
Measure: Mean (Standard Error); unit: cigarettes/day
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 24 | 18
cigarettes/day | 3.877 (1.179) | 4.29 (1.265)
Statistical Analysis 1: Comparison: Deep rTMS Active + Varenicline vs Deep rTMS Sham + Varenicline; Test type: Superiority; p = 0.98, Mixed Models Analysis; η2 = 0.02

5. Secondary Outcome: Minnesota Nicotine Withdrawal Scale (MNWS) Score
Description: This will be used to assess withdrawal symptoms. It is an 8 item scale and total scores range from 0 to 24. A higher score indicates more severe nicotine withdrawal.
Time Frame: 26 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 24 | 18
score on a scale | 8.291 (1.922) | 9.372 (2.107)
Statistical Analysis 1: Comparison: Deep rTMS Active + Varenicline vs Deep rTMS Sham + Varenicline; Test type: Superiority; p = 0.24, Mixed Models Analysis; η2 = 0.07

6. Secondary Outcome: Tiffany Questionnaire for Smoking Urges (T-QSU) Score
Description: This will be used to assess symptoms of craving/urges for tobacco. It is a 32 item scale and total scores range from 0 to 224. A higher score indicates more severe smoking craving/urges.
Time Frame: 26 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 24 | 18
score on a scale | 61.683 (9.624) | 73.236 (10.311)
Statistical Analysis 1: Comparison: Deep rTMS Active + Varenicline vs Deep rTMS Sham + Varenicline; Test type: Superiority; p = 0.26, Mixed Models Analysis; η2 = 0.17

7. Secondary Outcome: Point Prevalence Abstinence at the End of 4 Weeks
Description: Measured by self-report of smoking abstinence in the past 7 days and confirmed using plasma cotinine measurement.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 18 | 16
Participants
  Abstinent | 11 | 9
  Non-abstinent | 7 | 7

8. Secondary Outcome: Prolonged Abstinence From End of Treatment (Week 12) to End of Follow up (Week 26)
Description: Measured by self-report of smoking abstinence since the last visit and confirmed using plasma cotinine measurement.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 16 | 15
Participants
  Abstinent | 5 | 4
  Non-abstinent | 11 | 11

9. Secondary Outcome: Prolonged Abstinence With 2-week Grace Period at End of Follow up (Week 26)
Description: Measured by self-report of smoking abstinence since the last visit and confirmed using plasma cotinine measurement.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 16 | 15
Participants
  Abstinent | 5 | 4
  Non-abstinent | 11 | 11

10. Secondary Outcome: Continuous Abstinence at 6 Months
Description: Measured by self-report of smoking abstinence since the last visit and confirmed using plasma cotinine measurement.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
Number analyzed (Participants) | 16 | 15
Participants
  Abstinent | 5 | 4
  Non-abstinent | 11 | 11

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the study until end of study involvement (i.e., 6 months)
Arm/Group | Deep rTMS Active + Varenicline | Deep rTMS Sham + Varenicline
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/18
Other Adverse Events (participants affected / at risk) | 15/24 | 11/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep rTMS Active + Varenicline (N=24) | Deep rTMS Sham + Varenicline (N=18)
Nausea (Nervous system disorders) | 8 (8) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 6 (6)
Vivid Dreams (Product Issues) | 4 (4) | 2 (2)
Sleep Disturbances (Product Issues) | 2 (2) | 3 (3)
Diarrhea (Product Issues) | 2 (2) | 3 (3)
Fatigue (Product Issues) | 3 (3) | 2 (2)
Contispation/bloating (Product Issues) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Low Mood (Psychiatric disorders) | 2 (2) | 1 (1)
Dizzy (Nervous system disorders) | 1 (1) | 2 (2)
Leg pain/leg cramp (General disorders) | 2 (2) | 1 (1)
Nightmare (Product Issues) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Sore Throat (General disorders) | 1 (1) | 0 (0)
Runny Nose (General disorders) | 1 (1) | 0 (0)
Trouble Concentrating (General disorders) | 1 (1) | 0 (0)
Sweating (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0)
Joint Stiffness (General disorders) | 0 (0) | 1 (1)
Muscle Cramp (General disorders) | 0 (0) | 1 (1)
Phosphene (General disorders) | 1 (1) | 0 (0)
Face twitching (General disorders) | 1 (1) | 0 (0)
Acid Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Amoeba (General disorders) | 0 (0) | 1 (1)
Poor Memory (General disorders) | 0 (0) | 1 (1)
Dry Skin (General disorders) | 1 (1) | 0 (0)
Fentanyl Overdose (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT04083144/Prot_SAP_000.pdf